CLINICAL TRIAL: NCT02292966
Title: Impact of HCV Eradication on Neurocognitive Functions and CNS Metabolism: a Trial of Daclatasvir, Asunaprevir and Beclabuvir for Patients With HCV Genotype 1 Infection
Brief Title: Impact of HCV Treatment on Neurocognitive Functions and Brain Metabolism
Acronym: HEPCOG-II
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VHCRP1304
Record Dates: First submitted 2014-09-25; First posted 2014-11-18 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C; Hepatitis; Asunaprevir; Daclatasvir; Beclabuvir; Neurocognitive function; Brain metabolites; Direct acting antiviral therapy
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C; Hepatitis | interventions — daclatasvir; asunaprevir; 8-cyclohexyl-N-((dimethylamino)sulfonyl)-1,1a,2,12b-tetrahydro-11-methoxy-1a-((3-methyl-3,8-diazabicyclo(3.2.1)oct-8-yl)carbonyl)cycloprop(d)indolo(2,1-a)(2)benzazepine-5-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hepatitis C treatment (Experimental): 12 weeks of DCV/ASV/BCV therapy.
  Interventions: Drug: DCV/ASV/BCV

INTERVENTIONS:
Drug: DCV/ASV/BCV — Each participant will each receive daclatasvir (30mg), asunaprevir (200mg) and beclabuvir (75mg) in a fixed-dose combination oral tablet for twice daily administration with food.
  Other Names: Daclatasvir; Asunaprevir; Beclabuvir

SUMMARY:
The purpose of this study is to examine whether neurocognitive impairments experienced by patients with chronic hepatitis C virus (HCV) infection can be reversed by treating HCV, with a new combination of direct acting antiviral drugs (daclatasvir (DCV), asunaprevir (ASV) and beclabuvir (BCV)). The study will assess the effect of HCV on the central nervous system (CNS) by assessing neurocognitive function and brain injury prior to treatment, and comparing it to the end of treatment, and 4, 12 and 24 weeks after treatment.

DETAILED DESCRIPTION:
This study will evaluate the effect of DCV/ASV/BCV on neurocognitive functioning and brain metabolite concentrations in the frontal white matter and the basal ganglia in people with chronic HCV genotype 1 infection, through a comparison of baseline and post-treatment parameters.

This is an open label single arm multi-centre study. All participants will each receive daclatasvir (30mg), asunaprevir (200mg) and beclabuvir (75mg) in a fixed-dose combination oral tablet for twice daily administration with food.

Duration of treatment will be 12 weeks for all subjects followed by 24 weeks of observational follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65 years
* Chronic HCV infection as documented by positive HCV RNA at screening and positive HCV RNA or anti-HCV antibody at least 6 months prior to screening
* HCV genotype 1 - mixed subtype, indeterminate subtype or other variants of genotype 1 are permissible
* Non-advanced cirrhotic defined as FibroScan ≤9.6 kPA at screening
* HCV treatment naïve
* Seronegative for HIV and HBsAg
* HCV RNA level of ≥104 IU/mL (10,000 IU/mL)
* Body Mass Index (BMI) between 18 and 35 kg/m2
* Women of childbearing potential (WOCBP) must:

  i. Have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/mL or equivalent units of HCG) within 24 hours prior to the start of study drug ii. Not be breastfeeding iii. Agree to follow instructions for methods of contraception for the duration of the treatment and for five weeks post-treatment completion
* Men who are sexually active with WOCBP must agree to follow instructions for methods of contraception for the duration of the treatment and for 14 weeks post-treatment completion
* Sufficient proficiency in English to complete the neurocognitive assessment, as judged by the investigator

Exclusion Criteria:

Target disease

* Infected with HCV other than genotype 1

Medical history and concurrent diseases

* Current hazardous consumption of alcohol, defined by an AUDIT-C score ≥4 for men and ≥3 for women
* Illicit substance use, identified by urinary drug test at screening
* Past history of non HCV-related CNS disorder, including seizures and traumatic brain injury
* Currently on an SSRI or other neuropsychiatric therapy
* Liver or any other organ transplant other than cornea and hair
* Current or known history of cancer (except in situ carcinoma of the cervix or adequately treated basal or squamous cell carcinoma of the skin) within 5 years prior to enrolment
* Evidence of a medical condition contributing to chronic liver disease other than HCV (such, but not limited to: hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcohol liver disease)
* Any gastrointestinal disease or surgical procedure that may impact the absorption of study drug (subjects who have cholecystectomy are permitted to enter the study)
* Known history of coagulopathy including, but not limited to, hemophilia
* Uncontrolled diabetes defined as HbA1c >7% at screening
* Confirmed, uncontrolled hypertension (any screening systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg should be excluded unless discussed with the study medical monitor)
* Inability to tolerate oral medication
* Poor venous access
* Any other medical, psychiatric and/or social reason which, in the opinion of the investigator would make the subject inappropriate for the study

Physical and Laboratory Test Findings

* ALT ≥ 5 x ULN
* Total Bilirubin ≥ 34 µmol/L (≥ 2 mg/dl), unless subject has documented history of Gilbert's disease
* INR ≥ 1.3
* Albumin < 3.5 g/dL (35g/L)
* Platelets < 100 x 109 cells/L
* ANC < 0.75 x 109 cells/L
* Hemoglobin < 10 g/dL (100g/L)
* Creatinine clearance (CrCL) ≤ 50 mL/min
* Alpha fetoprotein (AFP) > 50ng/mL
* QTcF or QTcB > 580mSec
* Positive HBsAg, HIV-1 or HIV-2 Ab

Allergies and Adverse Drug Reaction

* History of hypersensitivity to drugs with a similar biochemical structure to DCV, ASV or BCV
* Any other criteria or know contraindication that would exclude the subject from receiving DCV, ASV or BCV Prohibited treatments and/or Therapies
* Exposure to any investigational drug or placebo within 4 weeks of study drug administration
* Refer to 5.5 for prohibited and/or restricted treatments during and post-treatment Sex and reproductive status
* Males and females who do not or are unable to meet the requirements outlined in Inclusion Criterias 9 and 10

Other Exclusion Criteria

* Prisoners or subjects who are involuntarily incarcerated
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g. infection disease) illness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-07; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Neurocognitive functioning | 36 weeks
  Mean change in neurocognitive functioning (global z-score representing overall neurocognitive performance across CogState, pegboard and colours trails)
Brain metabolite concentrations | 36 weeks
  Mean change in five absolute metabolite concentrations (NAA,Cho, Cr, mlo, glx)

SECONDARY OUTCOMES:
Neurocognitive functioning | 12 and 24 weeks
  Mean change in neurocognitive functioning (global z-score representing overall neurocognitive performance across CogState, pegboard and colours trails)
NAA metabolite concentration in the brain | 12 and 24 weeks
Cho metabolite concentration in the brain | 12 and 24 weeks
Cr metabolite concentration in the brain | 12 and 24 weeks
MLO metabolite concentration in the brain | 12 and 24 weeks
Glx metabolite concentration in the brain | 12 and 24 weeks
Change in neurocognitive functioning compared between subjects with and without sustained virological response (SVR) | 24 weeks
  Mean change in neurocognitive functioning (global z-score representing overall neurocognitive performance across CogState, pegboard and colours trails)
Change in brain metabolite concentrations compared between subjects with and without sustained virological response (SVR) | 24 weeks
  Mean change in absolute metabolite concentrations (NAA,Cho, Cr, mlo, glx)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Dore, BSc, MBBS, FRACP, MPH, PhD, Principal Investigator — Kirby Institute
Locations (2):
- Australia (2):
  - St Vincent's Hospital, Sydney, New South Wales
  - Westmead Hospital, Westmead, New South Wales